CLINICAL TRIAL: NCT04360096
Title: Inhaled ZYESAMI™ for the Treatment of Severe COVID-19
Brief Title: Inhaled ZYESAMI™ (Aviptadil Acetate) for the Treatment of Severe COVID-19
Acronym: AVICOVID-2
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: APR Applied Pharma Research s.a. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RLF-100_002
Record Dates: First submitted 2020-04-21; First posted 2020-04-24 (Actual); Last update posted 2023-02-03 (Actual); Status verified 2021-11

CONDITIONS: SARS-CoV 2; COVID; ARDS; ALI; Acute Lung Injury/Acute Respiratory Distress Syndrome (ARDS); Dyspnea
Keywords: Corona Virus; VIP; Aviptadil; Vasoactive Intestinal Polypeptide
MeSH Terms: conditions — Acute Lung Injury; Respiratory Distress Syndrome; Dyspnea | interventions — aviptadil

STUDY DESIGN:
Intervention Model Description: Multicenter Randomized Placebo-controlled Trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Only the study pharmacist will be aware of treatment assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (2):
- Severe COVID-19 ZYESAMI™ (Experimental): Patients with Severe COVID-19 to be treated with inhaled ZYESAMI™ (aviptadil) by mesh nebulizer 100μg 3x daily
  Interventions: Drug: ZYESAMI™ (aviptadil acetate); Device: Nebulized administration of ZYESAMI™ or Placebo
- Severe COVID-19 Placebo (Experimental): Patients with Severe COVID-19 to be treated with inhaled placebo 3x daily
  Interventions: Drug: Placebo; Device: Nebulized administration of ZYESAMI™ or Placebo

INTERVENTIONS:
Drug: ZYESAMI™ (aviptadil acetate) — Inhaled ZYESAMI™ (aviptadil acetate) 100μg 3x daily by mesh nebulizer
  Arms: Severe COVID-19 ZYESAMI™
Drug: Placebo — Normal Saline Inhalation
  Arms: Severe COVID-19 Placebo
Device: Nebulized administration of ZYESAMI™ or Placebo — Use of 510(k) cleared mesh nebulizer to deliver investigational product

SUMMARY:
Brief Summary:

SARS-CoV-2 virus infection is known to cause Lung Injury that begins as dyspnea and exercise intolerance, but may rapidly progress to Critical COVID-19 with Respiratory Failure and the need for noninvasive or mechanical ventilation. Mortality rates as high as 80% have been reported among those who require mechanical ventilation, despite best available intensive care.

Patients with severe COVID-19 by FDA definition who have not developed respiratory failure be treated with nebulized ZYESAMI™ (aviptadil acetate, a synthetic version of Vasoactive Intestinal Polypeptide (VIP)) 100 μg 3x daily plus Standard of Care vs. placebo + Standard of Care using an FDA 501(k) cleared mesh nebulizer.

The primary outcome will be progression in severity of COVID-19 (i.e. critical OR severe progressing to critical) over 28 days. Secondary outcomes will include blood oxygenation as measured by pulse oximetry, dyspnea, exercise tolerance, and levels of TNFα IL-6 and other cytokines.

DETAILED DESCRIPTION:
Detailed Description:

Attack of the Alveolar Type II (ATII) cell via its ACE2 surface receptor by the SARS-CoV-2 virus leads to respiratory failure, morbidity, and frequently mortality in COVID-19. There is no approved treatment that specifically targets the pulmonary injury. Vasoactive Intestinal Peptide (VIP) is known to target the VPAC1 receptor of the ATII cell and to protect that cell against all manner of injuries, including smoke inhalation, exposure to stomach acid, and exposure to infectious agents. VIP prevents apoptosis, blocks cytokines, lowers TNFα levels, reverses CD4/CD8 ratio, and reduces cough and dyspnea in nonclinical and clinical studies. Aviptadil acetate, a synthetic form of Vasoactive Intestinal Polypeptide (VIP) has been awarded FDA Orphan Drug Designation for the treatment of ARDS and Pulmonary Hypertension and EMEA Orphan Drug Designation for the treatment of ARDS and Sarcoid. ZYESAMI™ (Aviptadil) has been granted FDA Fast Track Designation for the treatment of ARDS/Acute Lung Injury in COVID-19.

The objective of this study is to identify patients severe COVID-19 who have not yet developed respiratory failure and to treat them with inhaled ZYESAMI™ in the hope of preventing progression to Critical COVID-19 with Respiratory Failure.

Nonclinical studies demonstrate that VIP is 70% concentrated in the lung, where it binds primarily to ATII cells. VIP prevents NMDA-induced caspase-3 activation in the lung, inhibits IL6 and TNFα production, protects against HCl-induced pulmonary edema, These and other effects have been observed in numerous animal model systems of lung injury in mice, rats, guinea pigs, sheep, swine, and dogs. In these models, Aviptadil restores barrier function at the endothelial/alveolar interface and thereby protects the lung and other organs from failure.

Both intravenous and inhalation preclinical toxicology and safety pharmacology have been performed in four species, with a six-month trial of inhaled Aviptadil in primates.

Aviptadil is approved for human use in the treatment of erectile dysfunction in Scandinavia and several European countries in co-formulation with phentolamine and has a demonstrated phase 2 safety in trials for Sarcoid, Pulmonary Fibrosis, and Bronchospasm. No adverse safety signals were seen in a phase I trial IV Aviptadil in ARDS. In that phase I trial, 8 patients with severe ARDS on mechanical ventilation were treated with ascending doses of VIP. Seven of the 8 patients were successfully extubated and were alive at the five-day timepoint. Six left the hospital and one died of an unrelated cardiac event.

A 60-day phase 2b/3 trial of IV Aviptadil (NCT 04311697) has recently completed enrollment and 28-day top-line safety data have been reported. No unanticipated serious adverse events were reported. The only adverse event that was statistically more frequent in Aviptadil-treated participants than among placebo-treated participants was mild to moderate diarrhea, which has not been reported as a frequent side-effect of inhaled Aviptadil (30% vs 1.5%; p< .001). Systemic hypotension was seen in both Aviptadil-treated and placebo-treated participants (25% vs 18.5%; P=NS).

Five GCP phase 2 trials of Aviptadil were conducted under European regulatory authority. Non GCP healthy volunteer studies have shown that i.v. infusion of Aviptadil is well tolerated with few adverse effects including alterations in blood pressure, heart rate, or ECG. In addition to published studies of human use, Aviptadil has been used on a compounded basis in certain ICUs for many years in the belief that it preserves life and restores function in pulmonary hypertension, ARDS, and Acute Lung Injury (ALI).

In this study, patients with severe COVID-19 by FDA definition who have not developed respiratory failure will be treated with nebulized ZYESAMI™ 100 μg in 1 cc normal saline 3x daily plus Standard of Care vs. placebo + Standard of Care using an FDA 501(k) cleared mesh nebulizer.

The primary outcome will be progression to in severity of COVID-19 (i.e. critical OR severe progressing to critical) over 28 days. Secondary outcomes will include blood oxygenation as measured by pulse oximetry, dyspnea, exercise tolerance, and levels of TNFα IL-6 and other cytokines.

ELIGIBILITY:
Inclusion criteria:

1. Severe COVID-19 , as defined by clinical signs indicative of severe systemic illness with COVID-19, being given oxygenation and meeting

   ONE of the following:

   Respiratory rate ≥ 30 per minute Heart rate ≥ 125 per minute SpO2 ≤ 93% on room air at sea level PaO2/FiO2 < 300 mmHg or SpO2/FiO2 < 315 mmHg
2. Positive test by standard RT-PCR assay or equivalent within last 7 days
3. Physician determination that patient is on SOC therapy, and will receive standard of care if patient progresses to Critical COVID-19, patient must be full CODE

Exclusion criteria:

1. Evidence of Critical COVID-19
2. Inability to utilize nebulized drugs, or history of bronchospasm with inhaled medications
3. Age <12 years;
4. Mean arterial pressure < 65 mm Hg after initial hospital stabilization,
5. Non-COVID-19 irreversible underlying condition with projected fatal course within 6 months or with high risk of mortality;
6. Immunosuppressive treatment for transplant or other diseases associated with high mortality;
7. Stage IV cancer or cancer on active treatment with chemotherapy immunotherapy or checkpoint inhibitors; acute renal failure or chronic renal insufficiency with GFR less than 30; CHF New York Heart Association class III or IV, new neurologic disorder in the last 3 months or chronic neurologic disorder or other that would impact on assessing the resolution of severe COVID-19 respiratory failure
8. Myocardial Infarction in previous six months or troponin >0.5
9. Recent history of venous thrombotic events (PE / DVT) within the last 3 months.
10. New diagnosis of atrial fibrillation within the last 3 months. Acceptable if greater than 3 months and well controlled in the opinion of the investigator
11. Watery diarrhea requiring replacement of 1 liter or more of iv fluids and electrolytes
12. Pregnancy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2021-02-15 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Progression to Respiratory Failure | 28 days
  Progression to Respiratory Failure is defined as the need for mechanical ventilation, non-invasive ventilation or high flow nasal oxygen

SECONDARY OUTCOMES:
Blood oxygenation | 28 days
  Blood PO2 as measured by pulse oximetry
RPD Dyspnea Scale | 28 days
  0 = no shortness of breath at all 0.5 = very, very slight shortness of breath
  1. = very mild shortness of breath
  2. = mild shortness of breath
  3. = moderate shortness of breath or breathing difficulty
  4. = somewhat severe shortness of breath
  5. = strong or hard breathing
  7 = severe shortness of breath or very hard breathing 8 9 = extremely severe shortness of breath 10 = shortness of breath so severe you need to stop the exercise or activity
Distance walked in six minutes | 28 days
  Distance walked in six minutes

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan C Javitt, MD, MPH, Study Chair — NeuroRx
Locations (13):
- United States (13):
  - St. Jude Medical Center, Fullerton, California
  - University of California - Irvine, Irvine, California
  - University of Miami Leonard M. Miller School of Medicine (UMMSM), Miami, Florida
  - Advent Health Research Institute, Orlando, Florida
  - Northwestern Medical Group, Winfield, Illinois
  - University of Louisville Hospital, Louisville, Kentucky
  - Great Plains Health, North Platte, Nebraska
  - University Medical Center, Las Vegas, Nevada
  - Holy Name Medical Center, Teaneck, New Jersey
  - Kettering Health Network, Kettering, Ohio
  - Doylestown Hospital, Doylestown, Pennsylvania
  - Self Regional Healthcare, Greenwood, South Carolina
  - University of Texas San Antonio Medical Arts and Research Center, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR

REFERENCES:
- See also: Pathogenesis of COVID-19 from a cell biologic perspective — https://erj.ersjournals.com/content/early/2020/03/17/13993003.00607-2020